CLINICAL TRIAL: NCT04652206
Title: An Open-label Phase Ib Prospective Clinical Trial to Investigate Safety, Tolerability and Maximum Tolerated Dose for SCO-101 in Combination With Gemcitabine and Nab-paclitaxel in Inoperable Pancreatic Cancer Patients.
Brief Title: Clinical Trial to Investigate Safety, Tolerability and MTD for SCO-101 in Combination With Gemcitabine and Nab-paclitaxel in Inoperable Pancreatic Cancer Patients.
Acronym: PANTAX-Ib
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scandion Oncology A/S (Industry)
Collaborators: Alcedis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCO101-002; 2020-002627-11 (EudraCT Number)
Record Dates: First submitted 2020-11-20; First posted 2020-12-03 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Locally Advanced Pancreatic Adenocarcinoma; Inoperable Disease; Localized Pancreatic Adenocarcinoma
Keywords: pancreatic; cancer; non-resectable; inoperable; pancreatic adenocarcinoma
MeSH Terms: conditions — Neoplasms | interventions — Gemcitabine; Taxes

STUDY DESIGN:
Intervention Model Description: Standard 3+3 dose escalation design to determine the Maximum Tolerated dose (MTD) of SCO-101 when administered in combination with gemcitabine and nab-paclitaxel, in patients with inoperable pancreatic cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCO-101 in combination with gemcitabine and nab-paclitaxel (Experimental): Patients receive escalating doses of SCO-101 in combination with the standard recommended dose of gemcitabine and nab-paclitaxel according to local clinical practice. Gemcintabine and nab-paclitaxel is the recommended treatment for the patient group.
  Starting dose of SCO-101 is 150 mg. Maximum dose tested is 350 mg. The dose is increased with 50 mg increments between each cohort.
  Interventions: Drug: SCO-101; Drug: Gemcitabine; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: SCO-101 — Oral tablets with a strength of 50 mg or 150 mg according to dose level (cohort). Administered for 6 consequtive days in a bi-weekly schedule in each treatment cycle. Treatment until disease progression.
Drug: Gemcitabine — Used according to marketing authorisation
Drug: Nab paclitaxel — Used according to marketing authorisation

SUMMARY:
An open-label dose escalating phase Ib study of SCO-101 in combination with gemcitabine and nab-paclitaxel. The primary objectives are to establish the safety profile and the MTD of SCO-101 when combined with gemcitabine and nab-paclitaxel. The starting dose of SCO-101 is 150 mg and the dose may be increased to a maximum of 350 mg.

DETAILED DESCRIPTION:
The study is an open-label dose escalating phase Ib study of SCO-101 in combination with gemcitabine and nab-paclitaxel. The primary objective is to establish the safety, tolerability and MTD of SCO-101 when combined with gemcitabine and nab-paclitaxel. Secondary objectives are efficacy and to establish PK parameters of SCO-101. The target indication is patients with inoperal pancreatic cancer who are to be treated with gemcitabine and nab-paclitaxel. The study is designed as a standard 3+3 dose escalation study with increasing doses of SCO-101 and a fixed dose (standard regimen) of gemcitabine and nab-paclitaxel. An interim report will be prepared once the last patient in the MTD cohort has completed one treatment cycle. Patients will continue treatment until disease progression to evaluate secondary objectives. One treatment Cycle is 28 days. The starting dose of SCO-101 is 150 mg 6 daily dosing in a bi-weekly schedule) and may be increased to a maximum of 350 mg (5 cohorts with 50 mg increments). A total of up to 18 patients are anticipated if dose escalation to the 5th cohort. Gemcitabine and nab-paclitaxel is administered according to local standard recommendations once weekly for three weeks followed by one weeks treatment holiday (dosing on day 6, day 13 and day 20). Patients may continue treatment until treatment progression.

ELIGIBILITY:
Inclusion Criteria:

Patients are required to meet all of the following criteria for enrollment into the study:

1. Ability to understand and willingness to provide written informed consent before any trial-related activities.
2. Age 18 years or older.
3. Histologically or cytologically verified pancreatic adenocarcinoma.
4. Inoperable localized, locally advanced or metastatic pancreatic cancer, not amenable for curatively intended treatment, in patients who are to be treated with gemcitabine and nab-paclitaxel.
5. Measurable or non-measurable disease determined by CT scan or MRI, according to RECIST 1.1.
6. Performance status of ECOG ≤ 2 and expected to tolerate the standard recommended (100%) gemcitabine and nab-paclitaxel dose.
7. Recovered to Grade 1 or less from prior surgery or acute toxicities of prior radiotherapy or treatment with cytotoxic or biologic agents.
8. ≥ 2 weeks must have elapsed since any prior surgery or radiotherapy.
9. Adequate conditions as evidenced by the following clinical laboratory values:

   * Absolute neutrophils count (ANC) ≥ 1.5 x 109/L
   * Haemoglobin ≥ 6.0 mmol/L
   * Platelets ≥ 100 x 109 /L
   * Alanine aminotransferase (ALT) ≤ 2.5 x ULN and aspartate aminotransferase (AST) ≤ 2.5 x ULN*
   * Total Serum bilirubin ≤ 1.0 ULN
   * Alkaline phosphatase ≤ 2.5 x ULN*
   * Creatinine ≤ 1.5 ULN
   * eGFR within normal limits
   * Adequate blood clothing function as defined by the International Normalized Ratio (INR) ≤ 1.2
10. Life expectancy longer than 3 months.
11. Sexually active males and females of child-producing potential must use highly effective contraception (intrauterine devices, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release)) for the study duration and at least 6 months after the last dose of study drug.
12. Signed informed consent. *AST is not mandatory. In case of known liver metastases with ALT and AST ≤ 5 x ULN and/or alkaline phosphatase ≤ 5 x ULN: Patients who do not conform to the transaminase and/or alkaline phosphatase inclusion criteria, but who by the PI are considered in good PS and otherwise eligible for inclusion, and where the transaminase and/or alkaline phosphatase levels are considered elevated due to other reasons than deteriorated lever capacity, may be considered for inclusion based on conferred agreement between PI and sponsor.

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from enrollment:

1. Concurrent chemotherapy, radiotherapy, or other investigational drug during study period.
2. Previous surgeries with resection of the complete stomach or greater part of small intestines (excluding the duodenum), whereby absorption of SCO-101 may be affected. Treatment with Creon or similar is allowed.
3. Difficulty in swallowing tablets.
4. CNS metastases requiring steroids.
5. Treatment with antibiotics for infections or with clinical symptoms of active infection. Patients showing symptoms of CoViD19 must be tested for active CoViD19 infection.
6. Known HIV positivity.
7. Known active hepatitis B or C.
8. Clinically significant (i.e. active) cardiovascular disease:

   * Stroke, Transient ischemic attack (TIA) or myocardial infarction within ≤ 6 months prior to day 1.
   * Unstable angina or NYHA Grade II or greater congestive heart failure (CHF).
   * Serious cardiac arrhythmia requiring medication.
9. Mental status, symptomatic epilepsy or other CNS disease where the investigator assesses the patient not fit for the clinical study.
10. Other medications or conditions that in the Investigator's opinion would contraindicate study participation of safety reasons or interfere with the interpretation of study results. Other severe medical conditions, including serious heart disease, unstable diabetes, uncontrolled hypercalcemia or previous organ transplants. Participation in another clinical trial with experimental medication within 30 days prior to registration.
11. Known hypersensitivity to gemcitabine and/or nab-paclitaxel.
12. Pregnant women or women who are breastfeeding.
13. Prior or present neuropathy > grade I (NCI-CTCAE v.5.0).
14. Curatively intended treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Through study completion, assessed up to 100 months
  Safety and tolerability by assessing the number, frequency, and severity of adverse events (AEs) collected from the time of first treatment until four weeks after end of treatment to evaluate safety of SCO-101 in combination with gemcitabine and nab-paclitaxel determined according to the Common Terminology Criteria for Adverse Events (NCI-CTCAE v.5.0).
Maximum Tolerated Dose | At the end of Cycle 1 (each cycle is 28 days)
  To determine the Maximum Tolerated Dose (MTD) of SCO-101 in combination with gemcitabine and nab-Paclitaxel by assessment of Dose Limiting Toxicities (DLT) to SCO-101.

SECONDARY OUTCOMES:
Objective Response Rate | Tumor assessment is performed every two treatment cycles (2 months), assessed up to 100 months.
  defined as CR and PR using the RECIST v. 1.1
Clinical Benefit Rate (CBR) | From benefit (CR, PR or SD > 16 weeks) to progression, assessed up to 100 months
  defined as the number of patients obtaining CR, PR, or SD > 16 weeks according to RECIST v.1.1.
Progression Free Survival (PFS) | From first dosing to progression, assessed up to 100 months
  defined as time in months from the date of first study treatment with SCO-101 to the date of disease progression or death from any cause, whichever comes first.
Overall Survival | through study completion, assessed up to 100 months
  defined as time in months from the date of first study treatment to the date of death
Pharmacokinetic profile | during the first 14 treatment days in the first treatment cycle.
  Pharmacokinetic profile of SCO-101 alone and in combination with gemcitabine and nab-paclitaxel

OTHER OUTCOMES:
Novel predictive biomarker feasibility | assessed from first administration to end of treatment, assessed up to 100 months.
  assessment of biomarkers from blood and tumor

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Odense Universitetshospital, Odense
- Germany (2):
  - Catholic Hospital Bochum - St. Josef-Hospital, Bochum
  - University Hospital Of Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No